CLINICAL TRIAL: NCT01862055
Title: Effect of Acute Preoperative Stress Assessed With Salivary Amylase on the Severity of Maternal Hypotension After Spinal Anesthesia for Planned Cesarean Section
Brief Title: Acute Preoperative Stress and Hypotension After Spinal Anesthesia. SAS for "Salivary Amylase and Stress "
Acronym: SAS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR 10010-NI09032; 2011-A00284-37 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2013-04-30; First posted 2013-05-24 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Planned Cesarean Section
Keywords: Stress; Anxiety; Cesarean Section; Spinal anesthesia; Hypotension
MeSH Terms: conditions — Anxiety Disorders; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Salivary samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SAS cohort: Consecutive patients undergoing planned cesarean section under spinal anesthesia

SUMMARY:
Spinal anesthesia is the technique of choice for planned cesarean section. It is associated with a high frequency of maternal hypotension. Hyperactivity of the sympathetic system assessed with the LF/HF ratio (heart rate variability analysis) predicts the severity of maternal hypotension after spinal anesthesia. Increased LF/HF ratio may be explained by maternal stress that can be measured with salivary amylase. The goal of this study is to assess the relationship between salivary amylase and severity of maternal hypotension after spinal anesthesia for planned cesarean section.

DETAILED DESCRIPTION:
Salivary amylase, heart rate variability, Spielberger state-trait inventory are assessed on the morning of surgery, on the surgical ward, and repeated in the operating room, before performing spinal anesthesia. Spinal anesthesia use hyperbaric bupivacaine (11 mg), sufentanil (5 µg) and morphine (100 µg). Prophylactic treatment of hypotension uses a continuous infusion of ephedrine (0.6 mg/ml) and phenylephrine (10 µg/ml). Rate of the continuous infusion is adapted to keep maternal systolic blood pressure between 95-105% of preinduction values. Total dose of ephedrine and phenylephrine infused from spinal anesthesia to delivery of the newborn is recorded (about 20 minutes for the estimated time frame). Association between stress markers and total dose of vasoactive drugs will be tested with the Spearman's correlation coefficient.

The study is observational. The subjects do receive a therapeutic intervention but the investigator does not assign patients to this intervention since this intervention is a routine care (spinal anesthesia for planned cesarian section) that would have been performed in the absence of the study.

ELIGIBILITY:
Pregnant women undergoing planned cesarean section under spinal anesthesia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women undergoing planned cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Severity of maternal hypotension assessed with the total dose of vasoactive drugs required to keep systolic blood pressure between 95-105% of preinduction values. | 20 minutes

SECONDARY OUTCOMES:
Salivary amylase activity | 20 minutes
  Measurement of amylase activity on a sample performed in the operating room, immediately before spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Dan Longrois, MD, PhD, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- HOPITAL BICHAT Claude Bernard, Paris, France